CLINICAL TRIAL: NCT06713876
Title: Long-term Outcomes of Patients Undergoing Extracorporeal Membrane Oxygenator-assisted Percutaneous Coronary Intervention
Brief Title: Long-term Outcomes of Patients Undergoing ECMO-assisted PCI
Status: Active, not recruiting | Type: Observational
Sponsor: Ling Tao, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Ling Tao, MD, PhD, Director of the Department of Cardiology, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: KY20242366-C-1
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Complex High-risk and Indicated Patients
Keywords: Percutaneous Coronary Intervention; ECMO; high-risk PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VA-ECMO-assisted PCI
  Interventions: Device: VA-ECMO-assisted PCI

INTERVENTIONS:
Device: VA-ECMO-assisted PCI — A total of 220 consecutive patients with VA-ECMO-assisted PCI will be enrolled. Data related to medical history, procedural characteristics, and outcomes were collected. Clinical follow-up will be conducted in the periprocedural and postoperative at 1 month, 1 year, 2 years, 3 years, 4 years, and 5 years.

SUMMARY:
Evidence regarding the long-term outcomes of patients undergoing Veno-arterial extracorporeal membrane oxygenator (VA-ECMO) assisted percutaneous coronary intervention (PCI) and the impact of the operator experience is limited.

The purpose of this retrospective single-center, observational registry in China is to investigate the long-term outcomes of patients undergoing VA-ECMO-assisted PCI and the impact of the operator experience.

DETAILED DESCRIPTION:
In the past four decades, there has been a widespread percutaneous coronary intervention (PCI) in coronary artery disease (CAD). Guidelines recommended that PCI is a reasonable option to improve survival, compared with medical therapy, in selected patients with low-to-medium anatomic complexity of CAD equally suitable for coronary artery bypass grafting (CABG); for complex and diffuse CAD, CABG was associated with a more significant clinical benefit. However, CABG is not always feasible due to patient preferences or the excess risk of perioperative morbidity and mortality. In selected patients with functionally significant multivessel disease (MVD) and LVEF ≤ 35% who are at high surgical risk or inoperable, PCI may be considered as an alternative to CABG. The recent 2024 European Society of Cardiology guidelines for the management of chronic coronary syndromes provided IIb B recommendation under such settings. However, such a subset of patients is considered at high risk for PCI complications due to the risk of hemodynamic collapse during balloon inflations or complex procedures.

Mechanical circulatory support (MCS) devices for elective high-risk PCI can provide hemodynamic support preventing hemodynamic failure during PCI. Several studies have suggested that intra aortic balloon pump (IABP) showed no significant benefits. Impella with a larger hemodynamic support also failed to demonstrate benefits, despite a tendency favoring the device. Venoarterial extracorporeal membrane oxygenation (VA -ECMO) is an alternative option for mechanical support, providing more extensive hemodynamic support in patients with potential or ongoing circulation failure. Initial reports on the use of VA-ECMO showed controversial results in the treatment of cardiogenic shock due to myocardial infarction. However, available evidence for the use of VA-ECMO in high-risk PCI has been restricted to retrospective small sizes; large-volume studies about the long-term outcome in this patient are limited.

ECMO requires a complex multidisciplinary approach and advanced technology. The potential benefits of hemodynamic support may be outweighed by the risk of device-associated complications, particularly bleeding and peripheral vascular events. Two studies have demonstrated that ECMO center experience may be associated with lower mortality in patients with cardiorespiratory failure. However, the relationship between operator experience and long-term outcomes post-VA-ECMO-assisted PCI in high-risk patients, and the ideal threshold to classify an operator as "experienced" have not been previously studied. Therefore, the aim of the present study was also to analyze the association between operator experience and one-year mortality post-VA-ECMO-assisted PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Coronary artery disease of the left main and/or multivessel disease
3. Combined with severely impaired left ventricular ejection fraction (LVEF), defined as LVEF ≤ 35% or decompensated heart failure
4. The heart team and the patient rejected CABG or OMT

Exclusion criteria were VA-ECMO support applied for cardiogenic shock or extracorporeal cardiopulmonary resuscitation (ECPR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated with VA-ECMO-assisted PCI
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
all-cause death | 1 year
  The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.

SECONDARY OUTCOMES:
cardiac death | 30 days, 1 year, 2 years, 3 years, 4 years, and 5 years
  The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.
myocardial infarction | 30 days, 1 year, 2 years, 3 years, 4 years, and 5 years
  The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.
stroke | 30 days, 1 year, 2 years, 3 years, 4 years, and 5 years
  Including ischemic stroke and hemorrhagic stroke. The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.
revascularization | 30 days, 1 year, 2 years, 3 years, 4 years, and 5 years
  Including target vessel revascularization and non-target vessel revascularization. The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.
rehospitalization | 30 days, 1 year, 2 years, 3 years, 4 years, and 5 years
  The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.
periprocedural complications | 30 days
  The outcome was defined according to the Mechanical Circulatory Support Academic Research Consortium definition.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D, Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng A, Wang B, Fu G, Li C, Liu Y, Li F, Wang Q, Yin Z, Gao H, Gao C, Tao L. Long-Term Outcomes of Patients Undergoing Extracorporeal Membrane Oxygenator-Assisted High-Risk Percutaneous Coronary Intervention. Catheter Cardiovasc Interv. 2025 Oct;106(4):2637-2644. doi: 10.1002/ccd.70098. Epub 2025 Aug 21. PMID 40842186